CLINICAL TRIAL: NCT06277843
Title: Development and Testing of a Low-cost and Reusable Thermal Jacket for Managing Preterm or Low-birth-weight Neonates in Bangladesh.
Brief Title: Low-Cost and Reusable Thermal Jacket for Managing Preterm or Low Birth Weight Neonates.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); Directorate General of Health Services (DGHS), Bangladesh (Unknown); Poeticgem International Ltd (Unknown); University of Dhaka (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-21131
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Preterm; Low Birthweight; Hypothermia Neonatal
Keywords: Preterm neonate; Low birthweight neonate; Kangaroo Mother Care; Thermal Jacket; Safety Trial
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Single arm non-randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal Jacket (Experimental)
  Interventions: Device: Thermal Jacket

INTERVENTIONS:
Device: Thermal Jacket — In the intervention group, the enrolled preterm or low birthweight eligible neonates gets the intervention (Thermal Jacket) as a supplement of Kangaroo Mother Care (KMC).

SUMMARY:
Globally, over 15 million neonates are born preterm each year. They account for approximately 30% of global neonatal deaths and 19% of total neonatal deaths in Bangladesh. They usually die because they cannot maintain normal temperature due to their weight, immature skin and underdeveloped thermal regulatory capacity of the brain.

Maintaining continuous KMC for at least 16-20 hours/day, is sometimes not feasible for mothers or caregivers. In addition, we also have the challenge of keeping preterm or LBW neonates warm during transportation.

The scientists at icddr,b, Johns Hopkins University, and George Mason University developed the re-usable thermal jacket for keeping preterm or low-birth-weight neonate warm. We propose to build on previous work by systematically testing the safety of the 'thermal jacket' among preterm or low birthweight (LBW) neonates.

Objective of this study is to conduct clinical safety trial of the thermal jacket to test whether the thermal jacket can retain euthermia of preterm or LBW neonates for 2 hours.

DETAILED DESCRIPTION:
We will equip a single arm trial with no control group design, in which every enrolled neonate will get the experimental therapy (thermal jacket) for this phase. A thermal jacket trial on a preterm or LBW neonate will be considered an event. An event will be considered a success if the neonate can maintain the body temperature in the euthermic range (36.5°C-37.5°C) using the thermal jacket for two hours. Thus, the failure event will be if the thermal jacket fails to maintain euthermia for neonates for two hours. Suppose, the neonate's body temperature drops below 36.5°C or rises above 37.5°C, the neonate will be monitored for maximum 5 minutes. If not recovered from the state, the neonate then immediately will be removed from the event for the appropriate management under the study's responsibility.

ELIGIBILITY:
Inclusion Criteria:

1. Neonate aged between 0-72 hours
2. Birthweight between 1800g to 2000g
3. No gross congenital anomaly
4. Normal heart 100-160 per minute
5. Capillary Refill Time ≤3 sec
6. Respiratory rate 30-59 per minute
7. Breaths comfortably (no chest indrawing, No gasping)
8. No sign of respiratory distress (respiratory rate within normal limit)
9. Pink in room air (without oxygen therapy)
10. H/O No prolonged or frequent apnea & no visible apnea during study enrolment
11. No major surgical problem

Exclusion Criteria:

1. In nasogastric tube
2. In oxygen therapy
3. In intravenous fluid

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Body temperature of preterm or low birthweight neonates and duration of time in euthermic range. | 2 hours per event
  Percentage of events maintained the body temperature in euthermic range among the enrolled preterm or low birthweight neonates.

CONTACTS AND LOCATIONS:
Overall Officials: Anisuddin Ahmed, MS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Bangladesh